CLINICAL TRIAL: NCT07297992
Title: The Effect of Simulation Training on Nursing Students' Perception, Myths and Attitudes of Dating Violence: A Randomized Controlled Study
Brief Title: The Effect of Simulation Training on Nursing Students' Perception, Myths and Attitudes of Dating Violence
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Makbule Tokur Kesgin, ASSOCIATE PROFESSOR, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AIBU-SBF-MTK-01
Record Dates: First submitted 2025-12-10; First posted 2025-12-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Nursing Students; Intimate Partner Violence (IPV)
Keywords: Intimate Partner Violence (IPV), high-fidelity simulation, Nursing Students, Flipped classroom, Randomised controlled trial

STUDY DESIGN:
Intervention Model Description: Arm 1 - Experimental: High-Fidelity Simulation-Based Education
  Arm 2 - Experimental: Flipped Classroom-Based Education
  Arm 3 - Control: Traditional Lecture-Based Education
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Fidelity Simulation-Based Education (Experimental)
  Interventions: Behavioral: High-Fidelity Simulation-Based Education
- Flipped Classroom-Based Education (Experimental)
  Interventions: Behavioral: Flipped Classroom-Based Education
- Control Grubu (No Intervention): A traditional lecture-based educational program on dating violence. The content is delivered through classroom lectures covering definitions, epidemiology, risk factors, myths, signs and symptoms, and reporting procedures related to dating violence. No simulation or flipped classroom components are included.

INTERVENTIONS:
Behavioral: High-Fidelity Simulation-Based Education — Nursing students in this group will receive an educational program on dating violence using high-fidelity simulation. Students will participate in realistic clinical scenario involving women exposed to dating violence, followed by debriefing and feedback sessions. The intervention is designed to improve students' recognition, assessment, and reporting of dating violence cases.
  Arms: High-Fidelity Simulation-Based Education
Behavioral: Flipped Classroom-Based Education — A flipped classroom educational program on dating violence. Students are provided with digital learning materials (videos, presentations, and readings) prior to class. During class sessions, students engage in discussions, case studies, and interactive activities focused on dating violence recognition, myths, and appropriate nursing care and reporting.
  Arms: Flipped Classroom-Based Education

SUMMARY:
Violence is a major global public health problem, causing approximately 1.5 million deaths each year. Dating violence, a common form of violence among young people, has serious consequences for women's and youths' physical and mental health, including mortality, chronic diseases, mental disorders, risky health behaviors, and substantial economic burden. As future healthcare providers, nursing students' myths, attitudes, and perceptions regarding dating violence can directly influence the quality and sensitivity of the care they deliver to survivors. Current literature mainly consists of descriptive studies focusing on nursing students' perceptions or attitudes toward dating violence, while experimental and structured educational interventions are limited.

This study aims to develop and evaluate an educational program supported by high-fidelity simulation and flipped learning to increase nursing students' awareness levels regarding dating violence, as well as to address their myths, attitudes, and perceptions. In the flipped learning component, students will review digital educational materials before class and actively participate in in-class activities; in the simulation component, students will engage in realistic scenarios involving dating violence cases to enhance their clinical readiness and care competencies. The study is designed to contribute to the prevention of dating violence by strengthening nursing students' knowledge, awareness, and professional responsibility in this field.

ELIGIBILITY:
Inclusion Criteria:

* To reside in the city center of Bartın
* To be a nursing student at Bartın University, Faculty of Health Sciences
* To have good Turkish communication skills
* To be 18 years of age or older
* To plan to live in Bartın for at least 6 months
* To be willing to participate in the study

Exclusion Criteria:

* To be enrolled at Bartın University as an exchange student during the active study period
* To have previously received simulation-based training on dating violence
* To participate in any other training program related to dating violence outside the study intervention
* To fail to respond to three or more contact attempts for the administration of post-training tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
Change in dating violence perception score | At this point, standardized scales will be used. Participants will be assessed with a pre-test before the training and a post-test after the training is completed. 2 mounth
  The Dating Violence Perceptions Scale will be used. The scale is a six-point Likert scale. Scale item scores are rated as follows: 1 = Strongly disagree, 2 = Disagree somewhat, 3 = Disagree slightly, 4 = Agree slightly, 5 = Agree somewhat, 6 = Strongly agree. The scale ranges from a minimum of 15 points to a maximum of 90 points. Higher scores on the scale indicate that the individual views dating violence as normal rather than abusive.
Change in dating violence myths belief score | At this point, a standardized scale will be used. Participants will be assessed with a pre-test before the training and a post-test after the training is completed. 2 mounth
  The Dating Violence Myths Scale will be used. The scale is a six-point Likert scale. Scale item scores are rated as follows: 1 = Strongly disagree, 2 = Disagree somewhat, 3 = Disagree a little, 4 = Agree a little, 5 = Agree somewhat, 6 = Strongly agree. The total score from the scale ranges from 9 to 54. A higher score on the scale indicates that the individual believes in dating violence myths.
Nursing Students' Perception and Understanding of Intimate Partner Violence Score | At this point, a standardized scale will be used. Participants will be assessed with a pre-test before the training and a post-test after the training is completed. 2 mounth
  The Scale of Nursing Students' Perceptions and Understanding of Intimate Partner Violence will be used. The scale item scores are based on a 5-point Likert-type rating system ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). The total score obtained from the scale ranges from 30 to 150. A higher score on the scale indicates a higher level of perception and understanding of intimate partner violence.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Büyüktopaç Büyüktopaç Çakıcı, Principal Investigator — Bartın Unıversity
Locations (1):
- Bartın University, Bartın, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Within 1-3 years after publication of the main study results, provided that participants have given their consent for data sharing.

REFERENCES:
- [Background] https://pubmed.ncbi.nlm.nih.gov/31793913/
- [Background] https://pubmed.ncbi.nlm.nih.gov/40168749/
- [Background] https://pubmed.ncbi.nlm.nih.gov/34085280/
- [Background] https://pubmed.ncbi.nlm.nih.gov/39705442/
- [Background] https://pubmed.ncbi.nlm.nih.gov/35272822/
- [Background] https://pubmed.ncbi.nlm.nih.gov/26753306/
- [Background] https://pubmed.ncbi.nlm.nih.gov/40290871/
- [Background] https://pubmed.ncbi.nlm.nih.gov/35779525/